CLINICAL TRIAL: NCT03925467
Title: Immediate Effects of Proximal and Distal Acupoints on the Radial Pressure Pulse-wave in Patients With Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Immediate Effects of Proximal and Distal Acupoints on the RPPW in Patients With KOA: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH108-REC2-033
Record Dates: First submitted 2019-04-21; First posted 2019-04-24 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; acupuncture; radial pressure pulse-wave; spectral energy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Three groups, pre-post intervention study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- proximal acupoints (Experimental): Acupuncture needles will be administered at proximal acupoints
  Interventions: Other: Acupuncture
- distal acupoints (Experimental): Acupuncture needles will be administered at distal acupoints
  Interventions: Other: Acupuncture
- sham acupoints (Placebo Comparator): Sham acupuncture needles will be administered in the abdominal sham acupoints.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Proximal acupoints: disposable acupuncture needles will be inserted into acupoints (GB34, SP9, EX-LE2) bilaterally for a depth of 10-30 mm.
  Distal acupoints: disposable acupuncture needles will be inserted into acupoints (LI11, HT3, TE10) bilaterally for a depth of 10-30 mm.
  Sham acupoints: Sham acupuncture needles will be administered into sham acupoints RN12, ST21.

SUMMARY:
Introduction: Knee osteoarthritis (KOA) is the most prevalent joint condition and is characterized by the progressive erosion of the articular cartilage. In TCM, Pulse Diagnosis has been one of the key diagnostic components in the clinical examinations. Modern pulse diagnosis studies have found that when the human body develops disease or is under pressure, the high frequency spectral energy (10-50Hz) will significantly change. Augmentation index (AIx) is related to the wave reflection of blood vessels. AIx can function as a useful index to reveal aging blood vessels. The experiment will use spectral energy and AIx as objective judgments about the efficacy of before-acupuncture and after-acupuncture treatment.

Method: This randomized controlled study will recruit 120 participants which will be allocated to 3 groups: Distal Acupoints, Proximal Acupoints and Sham Acupoints. Each group will have 40 participants to ensure a sufficient sample size can be attained for statistical analysis. Participants aged 20 or older with acute or chronic arthritis will be recruited when they meet the Clinical Classification Criteria for KOA, that is knee pain and three out of six symptoms can be found in clinical practices, as recommended by the American College of Rheumatology:(a) any gender aged 50 years or above;(b) have less than 30 mins of morning stiffness ; (c) crepitus on active motion; and (d)bony tenderness;(e)bony enlargement; and (f)no palpable warmth.Objective and subjective baseline assessments and outcome evaluations including VAS, The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and range of knee motion will be performed. The primary outcome will be the assessment of Spectral Energy and AIx of radial pressure pulse-wave in both wrists (Chun, Guan, and Chy pulse) using the Pulse Sphygmograph before and after the intervention. The secondary outcome involves evaluating VAS and range of knee motion.

Expected Outcome: The research findings can be clinical evidence regarding the effect of acupuncture KOA on radial artery. Moreover, the research will explore the immediate-effect difference between distal and proximal acupoints on KOA.

DETAILED DESCRIPTION:
Introduction: Knee osteoarthritis (KOA) is the most prevalent joint condition and is characterized by the progressive erosion of the articular cartilage. In TCM, Pulse Diagnosis has been one of the key diagnostic components in the clinical examinations. Modern pulse diagnosis studies have found that when the human body develops disease or is under pressure, the high frequency spectral energy (10-50Hz) will significantly change. Augmentation index (AIx) is related to the wave reflection of blood vessels. AIx can function as a useful index to reveal aging blood vessels. The experiment will use spectral energy and AIx as objective judgments about the efficacy of before-acupuncture and after-acupuncture treatment.

Method: This randomized controlled study will recruit 120 participants which will be allocated to 3 groups: Distal Acupoints, Proximal Acupoints and Sham Acupoints. Each group will have 40 participants to ensure a sufficient sample size can be attained for statistical analysis. Participants aged 20 or older with acute or chronic arthritis will be recruited when they meet the Clinical Classification Criteria for KOA, that is knee pain and three out of six symptoms can be found in clinical practices, as recommended by the American College of Rheumatology:(a) any gender aged 50 years or above;(b) have less than 30 mins of morning stiffness ; (c) crepitus on active motion; and (d)bony tenderness;(e)bony enlargement; and (f)no palpable warmth.Objective and subjective baseline assessments and outcome evaluations including VAS, The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and range of knee motion will be performed. The primary outcome will be the assessment of Spectral Energy and AIx of radial pressure pulse-wave in both wrists (Chun, Guan, and Chy pulse) using the Pulse Sphygmograph before and after the intervention. The secondary outcome involves evaluating VAS and range of knee motion.

Expected Outcome: The research findings can be clinical evidence regarding the effect of acupuncture KOA on radial artery. Moreover, the research will explore the immediate-effect difference between distal and proximal acupoints on KOA.

Other Information: The study will be conducted in China Medical University Hospital(Meide Medical Building) Acupuncture Department and Yiyuantang Chinese Medicine Clinic, Hsinchu City. Under the acupuncture of a qualified Chinese physician who has had at least 10 years of clinical experience, it is expected that the risk to the subject will not exceed the minimum risk. The investigators will begin data collection as soon as the approval of the Research Ethics Committee and the required equipment are available, and is expected to be completed within one year of the IRB approval.

ELIGIBILITY:
Inclusion Criteria:

Patients meet at least three out of the following six conditions:

* Any gender aged 50 years or above;
* Have less than 30 mins of morning stiffness;
* Crepitus on active motion;
* Bony tenderness;
* Bony enlargement;
* No palpable warmth.

Exclusion Criteria:

* Subjects who are unable to walk.
* Malignancy,
* Any acute medical condition,
* Poorly controlled diabetes or hypertension,
* A motor or sensory nerve defect,
* Blood clotting disease,
* Mental illness,
* Dementia,
* Mental retardation or other abnormal person on the organic mind.
* Subjects with intra-articular solid or hyaluronic acid injection in the past 3 months.
* Knee surgery,
* Knee trauma,
* Congenital knee deformation,
* Severe knee varus or valgus deformation,
* Endocrine,metabolic, infectious, inflammatory, secondary degenerative knee arthritis caused by problems with rheumatic immune diseases.
* Subjects who are hypersensitive to needles.
* Subjects who are unwilling to cooperate or sign the subject consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2020-03-24 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Radial Pressure Pulse-wave at cunkou (1) | 20 min before acupuncture
  Assessment of Radial Pressure Pulse-wave at cunkou ie at Cun, Guan & Chi of both hands before and after the intervention using Pulse Sphygmograph at 10 min before acupuncture.
Assessment of Radial Pressure Pulse-wave at cunkou (2) | 10 min after acupuncture
  Assessment of Radial Pressure Pulse-wave at cunkou ie at Cun, Guan & Chi of both hands before and after the intervention using Pulse Sphygmograph at 10 min after acupuncture.

SECONDARY OUTCOMES:
Range of knee motion | 1) 10 min before acupuncture; 2) within 20 min after needle removal
  Range of knee motion will be examined by a goniometer.
Visual analog scale (VAS) | 1) within 40 min before acupuncture; 2) within 20 min after needle removal
  The intensity of pain is measure using VAS for pain. It is incorporated into the questionnaire with a scale of 0 (no pain) to 10 (worst pain possible)
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | within 40 min before acupuncture
  A questionnaire developed to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, M.D.,PhD, Principal Investigator — China Medical University Hospital

IPD SHARING:
Plan to Share IPD: Undecided